CLINICAL TRIAL: NCT05716490
Title: Optimizing Closed Incision Negative Pressure Wound Therapy in Emergency Laparotomy: A Multi-arm Randomized Prospective Trial
Brief Title: Optimizing Closed Incision Negative Pressure Wound Therapy in Emergency Laparotomy
Acronym: OPTIWOUND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar do Tâmega e Sousa (Other)
Responsible Party: Principal Investigator, Marcelo José Maia Azevedo Costa, Principal investigator, general surgery resident, Centro Hospitalar do Tâmega e Sousa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 29/2022
Record Dates: First submitted 2023-01-28; First posted 2023-02-08 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Surgical Site Infection; Surgical Wound; Surgical Wound Infection; Surgical Complication; Surgical Wound Dehiscence; Surgical Wound Haemorrhage; Surgical Wound, Healed
Keywords: iNPWT; Incision negative pressure wound therapy; emergency laparotomy; general surgery; surgical site infection
MeSH Terms: conditions — Surgical Wound Infection; Surgical Wound; Surgical Wound Dehiscence

STUDY DESIGN:
Intervention Model Description: Patients are enrolled chronologically at the time of surgery into a slot of a previously randomized table with the 3 interventional arms
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard (Active Comparator): Control group which will cover surgical wound with conventional wound dressing
  Interventions: Other: Control group - standard wound dressing
- PICO (Experimental): Group that will use Pico® device for wound dressing
  Interventions: Device: Incisional negative pressure wound therapy
- PREVENA (Experimental): Group that will use Prevena® device for wound dressing
  Interventions: Device: Incisional negative pressure wound therapy

INTERVENTIONS:
Device: Incisional negative pressure wound therapy — Application of negative pressure wound therapy for prophylaxis of surgical site occurrences
  Arms: PICO; PREVENA
Other: Control group - standard wound dressing — Covering of surgical wound with standard wound dressing
  Arms: Standard

SUMMARY:
The purpose of this study is to find differences in rates of surgical site infections following emergency laparotomy with the use of two different incisional negative pressure wound therapy (iNPWT)devices.

DETAILED DESCRIPTION:
A multi-arm, randomized, single institution trial was conducted. All patients proposed for emergency laparotomy for different etiologies where considered eligible. Patients were enrolled following signature of informed consent.

Excluded from this group were patients with recent previous interventions (laparotomy or minimally invasive surgery), patients not wishing a iNPWT device or patients with specific contraindications to any device.

Later where excluded from the study patients on laparostomy, Intraoperative diagnosis of irreversible disease (Ex: Extensive mesenteric ischemia).

Following enrollment patients were randomized to 3 groups - control group with standard dressings; PICO group with Pico® (Smith & Nephew Inc, Andover, MA) dressing and Prevena group using Prevena® (KCI USA, Inc., San Antonio, TX) dressing.

Following admission the patients were monitored for surgical site occurrences and other complications by the investigation team until discharge. Subsequent 2 week post-operative evaluation (if patient had been discharged) was carried out in outpatient.

A final consultation was made 30 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* All patients proposed for emergency laparotomy

Exclusion Criteria:

* Contra-indication for iNPWT
* Irreversible disease diagnosis with expected short term mortality
* Need for a staged procedure

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | 30 days
  Surgical site infection following emergency laparotomy

SECONDARY OUTCOMES:
Surgical site occurrences | 30 days
  Seroma, hematoma, wound dehiscence

OTHER OUTCOMES:
Length of stay | 30 days
  post-operative length of stay
Reinterventions | 30 days
Adverse events related to devices | 30 days
Surgical complications | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo J Costa, MD, Principal Investigator — Centro Hospitalar do Tâmega e Sousa
Locations (1):
- Centro Hospitalar do Tâmega e Sousa, Penafiel, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No